CLINICAL TRIAL: NCT04195698
Title: A Phase 3b, Open-Label Treatment Extension Study of Upadacitinib for the Treatment of Adult Subjects With Moderate to Severe Atopic Dermatitis Who Completed Treatment in Study M16-046
Brief Title: Open-Label Extension Study of Upadacitinib in Adult Participants With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M19-850; 2019-001227-12 (EudraCT Number)
Record Dates: First submitted 2019-12-02; First posted 2019-12-12 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Upadacitinib; ABT-494; RINVOQ
MeSH Terms: conditions — Dermatitis, Atopic | interventions — upadacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Upadacitinib (Experimental): Participants will be administered with upadacitinib once daily (QD)
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Upadacitinib — Upadacitinib will be administered oral as tablet
  Other Names: ABT-494; RINVOQ

SUMMARY:
This is a study for adults (18-75 years) who have successfully completed treatment either with Dupilumab or with Upadacitinib in the study M16-046. At the end of M16-046, they have the option to receive Upadacitinib with a duration of 52 weeks beyond the timeframe of Study M16-046. There will be a 30 day follow-up visit after the treatment period is completed.

Main objective of this study is to assess long-term safety, tolerability and efficacy of upadacitinib in participants with moderate to severe atopic dermatitis who successfully completed treatment in the study M16-046.

ELIGIBILITY:
Inclusion Criteria:

* Participants should have successfully completed treatment in the M16-046 study, without meeting any permanent discontinuation criteria.
* Participant is judged to be in general good health (other than AD) as determined by the Principal Investigator and remains eligible as per the criteria for the study M16-046 to continue treatment in the long term extension study.

Exclusion Criteria:

* Requirement of prohibited medications during the study treatment or would interfere with appropriate assessment of atopic dermatitis lesions.
* Female participant who is pregnant, breastfeeding, or considering pregnancy during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (116):
- United States (33):
  - University of Arkansas for Medical Sciences /ID# 221021, Little Rock, Arkansas
  - Duplicate_First OC Dermatology Research Inc /ID# 218619, Fountain Valley, California
  - UCSF Fresno /ID# 218453, Fresno, California
  - California Allergy and Asthma Medical Group /ID# 218635, Los Angeles, California
  - Dermatology Research Associates /ID# 218637, Los Angeles, California
  - Dermatology Clinical Trials /ID# 218627, Newport Beach, California
  - Duplicate_UC Davis Health /ID# 218582, Sacramento, California
  - Ucsd /Id# 218629, San Diego, California
  - Clinical Science Institute /ID# 218632, Santa Monica, California
  - Miami Dermatology and Laser Institute /ID# 218664, Miami, Florida
  - Florida International Rsrch cr /ID# 218663, Miami, Florida
  - GCP Research /ID# 218665, St. Petersburg, Florida
  - Clinical Research Trials of Florida, Inc. /ID# 218438, Tampa, Florida
  - Georgia Pollens Clinical Research Centers, Inc /ID# 218441, Albany, Georgia
  - Medical Dermatology Associates of Chicago /ID# 218551, Chicago, Illinois
  - Sneeze, Wheeze, & Itch Associates, LLC /ID# 218552, Normal, Illinois
  - Dawes Fretzin, LLC /ID# 218478, Indianapolis, Indiana
  - Beacon Clinical Research, LLC /ID# 218636, Quincy, Massachusetts
  - Duplicate_Michigan Center for Research Company /ID# 218577, Clarkston, Michigan
  - Henry Ford Medical Center - New Center One /ID# 218575, Detroit, Michigan
  - Duplicate_Allergy, Asthma & Immunology Associates, PC /ID# 218548, Lincoln, Nebraska
  - Skin Specialists, PC /ID# 218549, Omaha, Nebraska
  - University Hospitals Case Medical Center /ID# 218574, Cleveland, Ohio
  - Southside Dermatology /ID# 218477, Tulsa, Oklahoma
  - Oregon Medical Research Center /ID# 218440, Portland, Oregon
  - Oregon Medical Research Center /ID# 218578, Portland, Oregon
  - Duplicate_Medical University of South Carolina /ID# 221072, Charleston, South Carolina
  - Clinical Research Solutions, LLC /ID# 218447, Jackson, Tennessee
  - Orion Clinical Research /ID# 218565, Austin, Texas
  - Sante Clinical Research /ID# 218911, Kerrville, Texas
  - Clinical Research Partners, LLC /ID# 218480, Richmond, Virginia
  - Duplicate_Premier Clinical Research /ID# 218583, Spokane, Washington
  - West Virginia Research Inst /ID# 218479, South Charleston, West Virginia
- Australia (5):
  - Holdsworth House Medical Practice /ID# 218755, Darlinghurst, New South Wales
  - The Skin Hospital /ID# 218753, Darlinghurst, New South Wales
  - Veracity Clinical Research /ID# 218754, Woolloongabba, Queensland
  - Sinclair Dermatology - Melbourne /ID# 218751, East Melbourne, Victoria
  - Burswood Dermatology /ID# 218752, Victoria Park, Western Australia
- Canada (10):
  - Kirk Barber Research, CA /ID# 218727, Calgary, Alberta
  - Duplicate_Dermatology Research Institute Inc. /ID# 218728, Calgary, Alberta
  - Dr. Chih-ho Hong Medical Inc. /ID# 218725, Surrey, British Columbia
  - Enverus Medical Research /ID# 218726, Surrey, British Columbia
  - Dr. Wei Jing Loo Medicine Prof /ID# 218722, London, Ontario
  - Duplicate_Lynderm Research Inc. /ID# 218723, Markham, Ontario
  - DermEdge Research Inc. /ID# 218721, Mississauga, Ontario
  - North York Research Inc /ID# 218729, Toronto, Ontario
  - Duplicate_K. Papp Clinical Research /ID# 218730, Waterloo, Ontario
  - Dre Angelique Gagne-Henley M.D. inc. /ID# 218724, Saint-Jérôme, Quebec
- Croatia (3):
  - DermaPlus - Poliklinika za dermatologiju i venerologiju /ID# 218377, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 218375, Zagreb, City of Zagreb
  - Naftalan - Specijalna bolnica za medicinsku rehabilitaciju /ID# 218376, Ivanić-Grad, Zagreb County
- Czechia (4):
  - Fakultni nemocnice Hradec Kralove /ID# 214176, Hradec Králové
  - Nemocnice Jihlava, prispevkova organizace /ID# 214178, Jihlava
  - Fakultni Nemocnice Ostrava /ID# 214177, Ostrava
  - Duplicate_Duplicate_Fakultni Nemocnice v Motole /ID# 214179, Prague
- Finland (3):
  - Keski-pohjanmaa Central Hospital /ID# 214630, Kokkola, Keski-Pohjanmaa
  - Duplicate_Oulun yliopistollinen sairaala /ID# 214628, Oulu, North Ostrobothnia
  - Mikkeli Central Hospital /ID# 214629, Mikkeli
- France (5):
  - AP-HM - Hopital de la Timone /ID# 218957, Marseille, Bouches-du-Rhone
  - Polyclinique Courlancy /ID# 218955, Reims, Marne
  - CHU de Nantes, Hotel Dieu -HME /ID# 218959, Nantes, Pays de la Loire Region
  - Hôpital Charles-Nicolle /ID# 218960, Rouen
  - CHU Toulouse - Hopital Larrey /ID# 218958, Toulouse
- Germany (6):
  - Dermatologische Mahlow /ID# 214225, Blankenfelde-Mahlow, Brandenburg
  - Duplicate_Klinikum Darmstadt GmbH /ID# 214224, Darmstadt, Hesse
  - Universitaetsklinikum Frankfurt /ID# 214223, Frankfurt am Main, Hesse
  - Duplicate_Universitaetsklinikum Muenster /ID# 214222, Munster, Lower Saxony
  - Medizinische Hochschule Hannover /ID# 214226, Hanover
  - Duplicate_Klinikum rechts der Isar - Technische Universitaet Muenchen /ID# 214221, Munich
- Hungary (3):
  - Oroshazi Korhaz /ID# 214986, Orosháza, Bekes County
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz /ID# 214984, Kaposvár, Somogy County
  - Uno Medical Trials Kft /ID# 214987, Budapest
- St Vincent's University Hospital /ID# 213558, Elm Park, Dublin, Ireland
- Israel (3):
  - Duplicate_HaEmek Medical Center /ID# 218520, Afula, Southern District
  - The Chaim Sheba Medical Center /ID# 218522, Ramat Gan, Tel Aviv
  - Rabin Medical Center /ID# 218521, Haifa
- Italy (4):
  - Istituto Clinico Humanitas /ID# 215727, Rozzano, Milano
  - Fondazione PTV Policlinico Tor Vergata /ID# 214093, Rome, Roma
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico /ID# 214095, Milan
  - Azienda Ospedaliero-Universitaria di Modena /ID# 214096, Modena
- Malaysia (6):
  - Hospital Sultan Ismail /ID# 218881, Johor Bahru, Johor
  - Hospital Pakar Sultanah Fatimah /ID# 218877, Muar town, Johor
  - Hospital Putrajaya /ID# 218880, Putrajaya, Putrajaya
  - Universiti Kebangsaan Malaysia (UKM) Medical Centre /ID# 218879, Kuala Lumpur, Selangor
  - Hospital Pulau Pinang /ID# 218878, George Town
  - University Malaya Med Ctr /ID# 218882, Kuala Lumpur
- Netherlands (4):
  - Bravis Ziekenhuis /ID# 218772, Bergen op Zoom, North Brabant
  - Duplicate_Erasmus Medisch Centrum /ID# 218770, Rotterdam, South Holland
  - Universitair Medisch Centrum Groningen /ID# 218775, Groningen
  - Universitair Medisch Centrum Utrecht /ID# 218771, Utrecht
- New Zealand (3):
  - Optimal Clinical Trials Ltd /ID# 218688, Grafotn, Auckland
  - Wellington Regional Hospital /ID# 218689, Newtown, Wellington Region
  - Clinical Trials New Zealand /ID# 218690, Hamilton
- Duplicate_Universitetssykehuset N-Norge, Tromso /ID# 214634, Tromsø, Troms, Norway
- Poland (5):
  - Duplicate_Pratia MCM Krakow /ID# 214303, Krakow, Lesser Poland Voivodeship
  - Klinika Ambroziak Sp. z o.o. /ID# 214301, Warsaw, Masovian Voivodeship
  - Duplicate_Duplicate_Royalderm Agnieszka Nawrocka /ID# 214302, Warsaw, Masovian Voivodeship
  - ClinicMed Daniluk, Nowak Sp.k. /ID# 214299, Bialystok, Podlaskie Voivodeship
  - Dermoklinika Centrum Medyczne s.c. /ID# 214300, Lodz, Łódź Voivodeship
- National University Hospital /ID# 219093, Singapore, Singapore
- Spain (6):
  - Duplicate_Hospital Universitario de Bellvitge /ID# 214257, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Dr. Negrin /ID# 214256, Las Palmas de Gran Canaria, Las Palmas
  - Hospital de Manises /ID# 214258, Manises, Valencia
  - Complejo Hospitalario Universitario de Pontevedra /ID# 214255, Pontevedra
  - Hospital Universitario Arnau Vilanova /ID# 214254, Valencia
  - Hospital Universitario y Politecnico La Fe /ID# 214252, Valencia
- Taiwan (4):
  - National Taiwan University Hospital /ID# 218917, Taipei City, Taipei
  - Chung Shan Medical University Hospital /ID# 218919, Taichung
  - China Medical University Hospital /ID# 218409, Taichung
  - Taipei Municipal Wan Fang Hospital /ID# 218918, Taipei
- Ukraine (2):
  - Kyiv City Clinical Skin and Venereal Hospital /ID# 218382, Kyiv, Kyivska Oblast
  - ME "Rivne Regional Dermatology and Venereology Dispensary" of RRC /ID# 218385, Rivne
- United Kingdom (4):
  - Victoria Hospital /ID# 213564, Kirkcaldy, Fife
  - Duplicate_The Royal Free London NHS Foundation Trust /ID# 213560, London, London, City of
  - NHS Greater Glasgow and Clyde /ID# 213561, Glasgow, Scotland
  - University Hospitals Sussex NHS Foundation Trust /ID# 213562, Worthing, West Sussex

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 475 participants were enrolled at 114 sites located in 22 countries (Australia, Canada, Croatia, Czechia, Finland, France, Germany, Hungary, Ireland, Israel, Italy, Malaysia, Netherlands, New Zealand, Norway, Poland, Singapore, Spain, Taiwan, Ukraine, United Kingdom, and the US).
Pre-assignment Details: Participants originally randomized to upadacitinib or dupilumab in Lead-In Study M16-046 and continued on into this Long-Term Extension Study M19-850.
  The ITT Population consists of all enrolled participants who received at least 1 dose of study drug in this study and is used for all efficacy analyses. The Safety Population is the same as the ITT Population and is used for all safety analyses.
Groups:
- DUPI 300mg to UPA 30mg: All participants in this study received upadacitinib 30 mg once a day (QD). Participants were grouped by previous treatment in Lead-In Study M16-046. Participants who received dupilumab (DUPI) in Lead-In Study M16-046 are included in the DUPI 300 mg Q2W/UPA 30 mg QD (DUPI/UPA) group.
- UPA 30mg to UPA 30mg: All participants in this study received upadacitinib 30 mg once a day (QD). Participants were grouped by previous treatment in Lead-In Study M16-046. Participants who received upadacitinib (UPA) in Lead-In Study M16-046 are included in the UPA 30 mg QD/UPA 30 mg QD (UPA/UPA) group.
Period: Overall Study
Arm/Group | DUPI 300mg to UPA 30mg | UPA 30mg to UPA 30mg
Started | 239 | 236
Completed | 214 | 197
Not Completed | 25 | 39
Not completed — Adverse Event | 4 | 11
Not completed — Withdrawal by Subject | 9 | 10
Not completed — Lost to Follow-up | 5 | 4
Not completed — Lack of Efficacy | 2 | 10
Not completed — Other | 5 | 4

BASELINE CHARACTERISTICS:
Population: The Baseline visit for this study was the Week 24 visit of Parent Study M16-046.
Groups:
- Total: Total of all reporting groups
Arm/Group | DUPI 300mg to UPA 30mg | UPA 30mg to UPA 30mg | Total
Number analyzed (Participants) | 239 | 236 | 475
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (12.90) | 36.1 (14.41) | 35.7 (13.66)
Age, Customized [Count of Participants; unit: Participants]
  Not Specified: < 40 years | 167 | 156 | 323
  Not Specified: ≥ 40 to < 65 years | 66 | 70 | 136
  Not Specified: ≥ 65 years | 6 | 10 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 104 | 204
  Male | 139 | 132 | 271
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 16 | 33
  Not Hispanic or Latino | 222 | 220 | 442
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 49 | 46 | 95
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 11 | 14 | 25
  White | 172 | 170 | 342
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: score on a scale] — EASI is a tool to measure the extent and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the percentage of skin affected, and the severity of eczema (scored as none [0], mild [1], moderate [2], or severe [3]) for redness, thickness, scratching, and lichenification are assessed. The EASI score is the sum of the scores for each region and ranges from 0 to 72, where higher scores represent worse disease.
  score on a scale | 3.26 (4.172) | 2.51 (4.274) | 2.89 (4.236)
Duration Since AD Diagnosis [Mean (Standard Deviation); unit: years] | 25.141 (13.6369) | 23.938 (14.9433) | 24.543 (14.2985)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: Treatment-emergent adverse events (TEAEs) are defined as any adverse events that begin or worsen in severity after initiation of upadacitinib during Lead-In Study M16-046 for the UPA/UPA arm or this Study M19-850 DUPI/UPA arm through 30 days following the last dose of upadacitinib.
Time Frame: UPA/UPA arm: BL visit in Lead-In M16-046 to last dose in Long-Term Extension M19-850 (median time on follow-up is 536 days); DUPI/UPA arm: BL visit in Long-Term Extension M19-850 to last dose plus a 30-day follow-up (median time on follow-up is 399 days).
Population: The Safety Population is the same as the ITT Population for this study. Safety summaries will include data collected from the first dose of updacitinib in Lead-In Study M16-046 or Study M19-850, whichever is earlier.
Measure: Count of Participants; unit: Participants
Arm/Group | DUPI 300mg to UPA 30mg | UPA 30mg to UPA 30mg
Number analyzed (Participants) | 239 | 236
Participants
  Any TEAE | 205 | 223
  TESAE | 14 | 17
  TEAE leading to discontinuation of study drug | 12 | 18

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events of Special Interest (AESI)
Description: Treatment-emergent adverse events were monitored throughout the study to identify any adverse events of special interest that may indicate a trend or risk to participants. AESIs are defined as any adverse events that begin or worsen in severity after initiation of upadacitinib during Study M16-046 for the UPA/UPA arm or Study M19-850 for the DUPI/UPA arm through 30 days following the last dose of upadacitinib.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | DUPI 300mg to UPA 30mg | UPA 30mg to UPA 30mg
Number analyzed (Participants) | 239 | 236
Participants
  Serious infections | 7 | 8
  Opportunistic infection excluding Tuberculosis and Herpes Zoster | 6 | 4
  Malignancy | 1 | 0
  Non-melanoma skin cancer (NMSC) | 0 | 0
  Malignancy excluding NMSC | 1 | 0
  Lymphoma | 0 | 0
  Hepatic disorder | 19 | 15
  Adjudicated gastrointestinal perforations | 0 | 0
  Anemia | 7 | 8
  Neutropenia | 10 | 8
  Lymphopenia | 4 | 5
  Herpes zoster | 26 | 25
  Creatine phosphokinase (CPK) elevation | 31 | 44
  Renal dysfunction | 0 | 0
  Active tuberculosis | 0 | 1
  Adjudicated MACE | 0 | 0
  Adjudicated VTE | 0 | 0

3. Primary Outcome: Percentage of Participants With Potentially Clinically Important (PCI) Laboratory Values as Assessed by the Investigator
Description: Clinical laboratory test values are considered PCI if they meet either the lower-limit or higher-limit PCI criteria defined in the categories below. Percentage of participants with PCI laboratory values are summarized for hematology and chemistry.
  The Number Analyzed is defined as the number of participants with at least one post-baseline value for the specific criteria.
  Post-baseline grade must also be more extreme (worse) than the baseline grade in order to be included in the count. If a participant does not have a baseline value then the participant would be counted in the numerator if the participant had at least one post-baseline.
  xULN = Times upper limit of the normal range.
Time Frame: From Baseline to 30 days following last dose of study drug (Week 52)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | DUPI 300mg to UPA 30mg | UPA 30mg to UPA 30mg
Number analyzed (Participants) | 239 | 236
percentage of participants
  Hemoglobin (G/L): Grade 3 (<80): number analyzed (Participants) | 238 | 236
  Hemoglobin (G/L): Grade 3 (<80) | 0 | 0.8
  Hemoglobin (G/L): Grade 3 or above: number analyzed (Participants) | 238 | 236
  Hemoglobin (G/L): Grade 3 or above | 0 | 0.8
  Platelets (10^9/L): Grade 3 (25-<50): number analyzed (Participants) | 238 | 236
  Platelets (10^9/L): Grade 3 (25-<50) | 0 | 0.4
  Platelets (10^9/L): Grade 4 (<25): number analyzed (Participants) | 238 | 236
  Platelets (10^9/L): Grade 4 (<25) | 0 | 0
  Platelets (10^9/L): Grade 3 or above: number analyzed (Participants) | 238 | 236
  Platelets (10^9/L): Grade 3 or above | 0 | 0.4
  Leukocytes (10^9/L): Grade 3 (1.0-<2.0): number analyzed (Participants) | 238 | 236
  Leukocytes (10^9/L): Grade 3 (1.0-<2.0) | 0 | 1.3
  Leukocytes (10^9/L): Grade 4 (<1.0): number analyzed (Participants) | 238 | 236
  Leukocytes (10^9/L): Grade 4 (<1.0) | 0 | 0
  Leukocytes (10^9/L): Grade 3 or above: number analyzed (Participants) | 238 | 236
  Leukocytes (10^9/L): Grade 3 or above | 0 | 1.3
  Neutrophils(10^9/L): Grade 3 (0.5-<1.0): number analyzed (Participants) | 238 | 236
  Neutrophils(10^9/L): Grade 3 (0.5-<1.0) | 2.5 | 3.4
  Neutrophils(10^9/L): Grade 4 (<0.5): number analyzed (Participants) | 238 | 236
  Neutrophils(10^9/L): Grade 4 (<0.5) | 0.4 | 0.4
  Neutrophils(10^9/L): Grade 3 or above: number analyzed (Participants) | 238 | 236
  Neutrophils(10^9/L): Grade 3 or above | 2.9 | 3.8
  Lymphocytes(10^9/L): Grade 3 (0.2-<0.5): number analyzed (Participants) | 238 | 236
  Lymphocytes(10^9/L): Grade 3 (0.2-<0.5) | 0.8 | 3.4
  Lymphocytes(10^9/L): Grade 4 (<0.2): number analyzed (Participants) | 238 | 236
  Lymphocytes(10^9/L): Grade 4 (<0.2) | 0 | 0.4
  Lymphocytes(10^9/L): Grade 3 or above: number analyzed (Participants) | 238 | 236
  Lymphocytes(10^9/L): Grade 3 or above | 0.8 | 3.8
  Alanine Aminotransferase (U/L): Grade 3 (>5.0-20.0 xULN): number analyzed (Participants) | 238 | 236
  Alanine Aminotransferase (U/L): Grade 3 (>5.0-20.0 xULN) | 0.4 | 0.4
  Alanine Aminotransferase (U/L): Grade 4 (>20.0 xULN): number analyzed (Participants) | 238 | 236
  Alanine Aminotransferase (U/L): Grade 4 (>20.0 xULN) | 0 | 0
  Alanine Aminotransferase (U/L): Grade 3 or above: number analyzed (Participants) | 238 | 236
  Alanine Aminotransferase (U/L): Grade 3 or above | 0.4 | 0.4
  Aspartate Aminotransferase (U/L): Grade 3 (>5.0-20.0 xULN): number analyzed (Participants) | 238 | 236
  Aspartate Aminotransferase (U/L): Grade 3 (>5.0-20.0 xULN) | 0 | 1.3
  Aspartate Aminotransferase (U/L): Grade 4 (>20.0 xULN): number analyzed (Participants) | 238 | 236
  Aspartate Aminotransferase (U/L): Grade 4 (>20.0 xULN) | 0 | 0
  Aspartate Aminotransferase (U/L): Grade 3 or above: number analyzed (Participants) | 238 | 236
  Aspartate Aminotransferase (U/L): Grade 3 or above | 0 | 1.3
  Alkaline Phosphatase (U/L): Grade 3 (>5.0-20.0 xULN): number analyzed (Participants) | 238 | 236
  Alkaline Phosphatase (U/L): Grade 3 (>5.0-20.0 xULN) | 0 | 0
  Alkaline Phosphatase (U/L): Grade 4 (>20.0 xULN): number analyzed (Participants) | 238 | 236
  Alkaline Phosphatase (U/L): Grade 4 (>20.0 xULN) | 0 | 0
  Alkaline Phosphatase (U/L): Grade 3 or above: number analyzed (Participants) | 238 | 236
  Alkaline Phosphatase (U/L): Grade 3 or above | 0 | 0
  Creatine Kinase (U/L): Grade 3 (>5.0-10.0 xULN): number analyzed (Participants) | 238 | 236
  Creatine Kinase (U/L): Grade 3 (>5.0-10.0 xULN) | 4.2 | 8.1
  Creatine Kinase (U/L): Grade 4 (>10.0 xULN): number analyzed (Participants) | 238 | 236
  Creatine Kinase (U/L): Grade 4 (>10.0 xULN) | 3.8 | 5.1
  Creatine Kinase (U/L): Grade 3 or above: number analyzed (Participants) | 238 | 236
  Creatine Kinase (U/L): Grade 3 or above | 8.0 | 13.1
  Creatinine (UMOL/L): Grade 3 (>3.0-6.0 xULN OR >3.0 xBaseline): number analyzed (Participants) | 238 | 236
  Creatinine (UMOL/L): Grade 3 (>3.0-6.0 xULN OR >3.0 xBaseline) | 0 | 0.8
  Creatinine (UMOL/L): Grade 4 (>6.0 xULN): number analyzed (Participants) | 238 | 236
  Creatinine (UMOL/L): Grade 4 (>6.0 xULN) | 0 | 0.4
  Creatinine (UMOL/L): Grade 3 or above: number analyzed (Participants) | 238 | 236
  Creatinine (UMOL/L): Grade 3 or above | 0 | 1.3
  Phosphate (MMOL/L): Grade 3 (0.3-<0.6): number analyzed (Participants) | 238 | 236
  Phosphate (MMOL/L): Grade 3 (0.3-<0.6) | 1.7 | 1.3
  Phosphate (MMOL/L): Grade 4 (<0.3): number analyzed (Participants) | 238 | 236
  Phosphate (MMOL/L): Grade 4 (<0.3) | 0 | 0
  Phosphate (MMOL/L): Grade 3 or above: number analyzed (Participants) | 238 | 236
  Phosphate (MMOL/L): Grade 3 or above | 1.7 | 1.3
  Calcium Hyper (MMOL/L): Grade 3 (>3.1-3.4): number analyzed (Participants) | 238 | 236
  Calcium Hyper (MMOL/L): Grade 3 (>3.1-3.4) | 0 | 0.4
  Calcium Hyper (MMOL/L): Grade 4 (>3.4): number analyzed (Participants) | 238 | 236
  Calcium Hyper (MMOL/L): Grade 4 (>3.4) | 0 | 0
  Calcium Hyper (MMOL/L): Grade 3 or above: number analyzed (Participants) | 238 | 236
  Calcium Hyper (MMOL/L): Grade 3 or above | 0 | 0.4
  Calcium Hypo (MMOL/L): Grade 3 (1.5-<1.75): number analyzed (Participants) | 238 | 236
  Calcium Hypo (MMOL/L): Grade 3 (1.5-<1.75) | 0 | 0
  Calcium Hypo (MMOL/L): Grade 4 (<1.5): number analyzed (Participants) | 238 | 236
  Calcium Hypo (MMOL/L): Grade 4 (<1.5) | 0 | 0.4
  Calcium Hypo (MMOL/L): Grade 3 or above: number analyzed (Participants) | 238 | 236
  Calcium Hypo (MMOL/L): Grade 3 or above | 0 | 0.4
  Sodium Hyper (MMOL/L): Grade 3 (>155-160): number analyzed (Participants) | 212 | 236
  Sodium Hyper (MMOL/L): Grade 3 (>155-160) | 0.5 | 0
  Sodium Hyper (MMOL/L): Grade 4 (>160): number analyzed (Participants) | 212 | 236
  Sodium Hyper (MMOL/L): Grade 4 (>160) | 0 | 0
  Sodium Hyper (MMOL/L): Grade 3 or above: number analyzed (Participants) | 212 | 236
  Sodium Hyper (MMOL/L): Grade 3 or above | 0.5 | 0
  Sodium Hypo (MMOL/L): Grade 3 (120-<130): number analyzed (Participants) | 212 | 236
  Sodium Hypo (MMOL/L): Grade 3 (120-<130) | 0 | 0.4
  Sodium Hypo (MMOL/L): Grade 4 (<120): number analyzed (Participants) | 212 | 236
  Sodium Hypo (MMOL/L): Grade 4 (<120) | 0 | 0
  Sodium Hypo (MMOL/L): Grade 3 or above: number analyzed (Participants) | 212 | 236
  Sodium Hypo (MMOL/L): Grade 3 or above | 0 | 0.4
  Potassium Hyper (MMOL/L): Grade 3 (>6.0-7.0): number analyzed (Participants) | 212 | 236
  Potassium Hyper (MMOL/L): Grade 3 (>6.0-7.0) | 0 | 0
  Potassium Hyper (MMOL/L): Grade 4 (>7.0): number analyzed (Participants) | 212 | 236
  Potassium Hyper (MMOL/L): Grade 4 (>7.0) | 0 | 0
  Potassium Hyper (MMOL/L): Grade 3 or above: number analyzed (Participants) | 212 | 236
  Potassium Hyper (MMOL/L): Grade 3 or above | 0 | 0
  Potassium Hypo (MMOL/L): Grade 3 (2.5-<3.0): number analyzed (Participants) | 212 | 236
  Potassium Hypo (MMOL/L): Grade 3 (2.5-<3.0) | 0 | 0
  Potassium Hypo (MMOL/L): Grade 4 (<2.5): number analyzed (Participants) | 212 | 236
  Potassium Hypo (MMOL/L): Grade 4 (<2.5) | 0 | 0
  Potassium Hypo (MMOL/L): Grade 3 or above: number analyzed (Participants) | 212 | 236
  Potassium Hypo (MMOL/L): Grade 3 or above | 0 | 0
  Glucose Hyper (MMOL/L): Grade 3 (>13.9-27.8): number analyzed (Participants) | 238 | 236
  Glucose Hyper (MMOL/L): Grade 3 (>13.9-27.8) | 1.3 | 0.4
  Glucose Hyper (MMOL/L): Grade 4 (>27.8): number analyzed (Participants) | 238 | 236
  Glucose Hyper (MMOL/L): Grade 4 (>27.8) | 0 | 0
  Glucose Hyper (MMOL/L): Grade 3 or above: number analyzed (Participants) | 238 | 236
  Glucose Hyper (MMOL/L): Grade 3 or above | 1.3 | 0.4
  Glucose Hypo (MMOL/L): Grade 3 (1.7-<2.2): number analyzed (Participants) | 238 | 236
  Glucose Hypo (MMOL/L): Grade 3 (1.7-<2.2) | 0 | 0
  Glucose Hypo (MMOL/L): Grade 4 (<1.7): number analyzed (Participants) | 238 | 236
  Glucose Hypo (MMOL/L): Grade 4 (<1.7) | 0 | 0
  Glucose Hypo (MMOL/L): Grade 3 or above: number analyzed (Participants) | 238 | 236
  Glucose Hypo (MMOL/L): Grade 3 or above | 0 | 0
  Albumin (G/L): Grade 3 (<20): number analyzed (Participants) | 238 | 236
  Albumin (G/L): Grade 3 (<20) | 0 | 0
  Albumin (G/L): Grade 3 or above: number analyzed (Participants) | 238 | 236
  Albumin (G/L): Grade 3 or above | 0 | 0
  Cholesterol (MMOL/L): Grade 3 (10.34<-12.92): number analyzed (Participants) | 238 | 236
  Cholesterol (MMOL/L): Grade 3 (10.34<-12.92) | 1.3 | 0
  Cholesterol (MMOL/L): Grade 4 (>12.92): number analyzed (Participants) | 238 | 236
  Cholesterol (MMOL/L): Grade 4 (>12.92) | 0 | 0
  Cholesterol (MMOL/L): Grade 3 or above: number analyzed (Participants) | 238 | 236
  Cholesterol (MMOL/L): Grade 3 or above | 1.3 | 0
  Triglycerides (MMOL/L): Grade 3 (>5.7-11.4): number analyzed (Participants) | 238 | 236
  Triglycerides (MMOL/L): Grade 3 (>5.7-11.4) | 3.4 | 5.1
  Triglycerides (MMOL/L): Grade 4 (>11.4): number analyzed (Participants) | 238 | 236
  Triglycerides (MMOL/L): Grade 4 (>11.4) | 0 | 0
  Triglycerides (MMOL/L): Grade 3 or above: number analyzed (Participants) | 238 | 236
  Triglycerides (MMOL/L): Grade 3 or above | 3.4 | 5.1

4. Primary Outcome: Percentage of Participants With Potentially Clinically Important (PCI) Vital Sign Measurements and Physical Examination Findings as Assessed by the Investigator
Description: PCI post-baseline vital sign values are summarized for categories: systolic and diastolic blood pressures [sitting], pulse rate [sitting], and weight. Only those categories where at least 1 person had a non-PCI value at Baseline and met the PCI criterion at least once during post-baseline are reported.
  The Number Analyzed is defined as the number of participants with at least one post-baseline value for the specific criteria.
  Post-baseline grade must also be more extreme (worse) than the baseline grade in order to be included in the count. If a participant does not have a baseline value then the participant would be counted in the numerator if the participant had at least one post-baseline.
Time Frame: From Baseline to 30 days following last dose of study drug (Week 52)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | DUPI 300mg to UPA 30mg | UPA 30mg to UPA 30mg
Number analyzed (Participants) | 239 | 236
percentage of participants
  Sitting Systolic Blood Pressure (MMHG): ≤90 and ≥20 Decrease: number analyzed (Participants) | 238 | 236
  Sitting Systolic Blood Pressure (MMHG): ≤90 and ≥20 Decrease | 0.4 | 0.8
  Sitting Systolic Blood Pressure (MMHG): ≥160 and ≥20 Increase: number analyzed (Participants) | 238 | 236
  Sitting Systolic Blood Pressure (MMHG): ≥160 and ≥20 Increase | 2.5 | 5.5
  Sitting Diastolic Blood Pressure (MMHG): ≤50 and ≥10 Decrease: number analyzed (Participants) | 238 | 236
  Sitting Diastolic Blood Pressure (MMHG): ≤50 and ≥10 Decrease | 0.4 | 1.3
  Sitting Diastolic Blood Pressure (MMHG): ≥100 and ≥10 Increase: number analyzed (Participants) | 238 | 236
  Sitting Diastolic Blood Pressure (MMHG): ≥100 and ≥10 Increase | 2.1 | 9.3
  Sitting Pulse Rate (BEATS/MIN): ≤50 and ≥15 Decrease: number analyzed (Participants) | 238 | 236
  Sitting Pulse Rate (BEATS/MIN): ≤50 and ≥15 Decrease | 1.7 | 4.7
  Sitting Pulse Rate (BEATS/MIN): ≥120 and ≥15 Increase: number analyzed (Participants) | 238 | 236
  Sitting Pulse Rate (BEATS/MIN): ≥120 and ≥15 Increase | 0 | 2.1
  Weight (KG): >7% Decrease: number analyzed (Participants) | 236 | 236
  Weight (KG): >7% Decrease | 5.5 | 7.6
  Weight (KG): >7% Increase: number analyzed (Participants) | 236 | 236
  Weight (KG): >7% Increase | 22.5 | 39.0

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include treatment-emergent events reported from the time of informed consent to end of study in M19-850 (52 weeks of treatment plus a 30 day follow-up after last dose). The median time on follow-up was 398 & 399 days for UPA/UPA & DUPI/UPA, respectively.
Groups:
- Total: All participants in this study received upadacitinib 30 mg once a day (QD). Participants were grouped by previous treatment in Lead-In Study M16-046. Participants who received upadacitinib (UPA) in Lead-In Study M16-046 are included in the UPA 30 mg QD/UPA 30 mg QD (UPA/UPA) group and participants who received dupilumab (DUPI) in Lead-In Study M16-046 are included in the DUPI 300 mg Q2W/UPA 30 mg QD (DUPI/UPA) group.
Arm/Group | UPA 30mg to UPA 30mg | DUPI 300mg to UPA 30mg | Total
All-Cause Mortality (participants affected / at risk) | 1/236 | 0/239 | 1/475
Serious Adverse Events (participants affected / at risk) | 13/236 | 14/239 | 27/475
Other Adverse Events (participants affected / at risk) | 154/236 | 149/239 | 303/475
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UPA 30mg to UPA 30mg (N=236) | DUPI 300mg to UPA 30mg (N=239) | Total (N=475)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
FOOD ALLERGY (Immune system disorders) | 1 (2) | 0 (0) | 1 (2)
ABSCESS JAW (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
BONE TUBERCULOSIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
BULLOUS IMPETIGO (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
COVID-19 PNEUMONIA (Infections and infestations) | 3 (3) | 0 (0) | 3 (3)
ECZEMA HERPETICUM (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
ERYSIPELAS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
PERICHONDRITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
PILONIDAL DISEASE (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
HAEMOGLOBIN DECREASED (Investigations) | 1 (1) | 0 (0) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 2 (2)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
ADNEXAL TORSION (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
ENDOMETRIOSIS (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
ABORTION INDUCED (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
ESSENTIAL HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UPA 30mg to UPA 30mg (N=236) | DUPI 300mg to UPA 30mg (N=239) | Total (N=475)
COVID-19 (Infections and infestations) | 31 (34) | 32 (34) | 63 (68)
HERPES SIMPLEX (Infections and infestations) | 12 (13) | 8 (10) | 20 (23)
HERPES ZOSTER (Infections and infestations) | 19 (20) | 25 (25) | 44 (45)
NASOPHARYNGITIS (Infections and infestations) | 15 (23) | 26 (35) | 41 (58)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 12 (13) | 14 (24) | 26 (37)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 35 (47) | 31 (42) | 66 (89)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 13 (14) | 1 (1) | 14 (15)
HEADACHE (Nervous system disorders) | 15 (22) | 14 (16) | 29 (38)
ACNE (Skin and subcutaneous tissue disorders) | 54 (65) | 49 (53) | 103 (118)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 45 (61) | 30 (48) | 75 (109)
ECZEMA (Skin and subcutaneous tissue disorders) | 14 (32) | 13 (17) | 27 (49)
HYPERTENSION (Vascular disorders) | 14 (14) | 4 (4) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-01-07): https://cdn.clinicaltrials.gov/large-docs/98/NCT04195698/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT04195698/SAP_001.pdf